CLINICAL TRIAL: NCT03906331
Title: Expanded Access for the Treatment of Cancers With Rearranged During Transfection (RET) Activation
Status: Approved for marketing | Type: Expanded Access
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Other Study IDs: 17494; Selpercatinib EAP (Other: Loxo Oncology, Inc.); J2G-OX-Y001 (Other: Eli Lilly and Company)
Record Dates: First submitted 2019-04-04; First posted 2019-04-08 (Actual); Last update posted 2025-01-17 (Actual); Status verified 2024-12

CONDITIONS: Non Small Cell Lung Cancer; Medullary Thyroid Cancer; Colon Cancer; Breast Cancer; Pancreatic Cancer; Papillary Thyroid Cancer; Other Solid Tumors With Evidence of Activating RET Alteration
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Carcinoma, Medullary; Colonic Neoplasms; Breast Neoplasms; Pancreatic Neoplasms; Thyroid Cancer, Papillary | interventions — selpercatinib

STUDY DESIGN:
Expanded Access Types: Individual

INTERVENTIONS:
Drug: Selpercatinib — Open-label expanded access
  Other Names: LOXO-292; LY3527723

SUMMARY:
Expanded access for participants with cancer with RET activation who are ineligible for an ongoing selpercatinib (also known as LOXO-292) clinical trial or have other considerations that prevent access to selpercatinib through an existing clinical trial.

The treating physician/investigator contacts Lilly when, based on their medical opinion, a patient meets the criteria for inclusion in the expanded access program.

DETAILED DESCRIPTION:
N/A for expanded access

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of cancer with RET activation, who are not eligible for an ongoing selpercatinib clinical trial and are medically suitable for treatment with selpercatinib
* Have progressed or are intolerant to standard therapy, or no standard therapy option exists, or in the opinion of the investigator, are unlikely to derive significant clinical benefit from standard therapy
* Have adequate organ function

Exclusion Criteria:

* Currently enrolled in an ongoing clinical study of selpercatinib or another RET inhibitor
* Clinically significant active cardiovascular disease or history of myocardial infarction within 6 months prior to study treatment; ongoing cardiomyopathy; or current prolongation of the QT interval corrected for heart rate using Fridericia's formula (QTcF) interval greater than 470 milliseconds

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult

CONTACTS AND LOCATIONS:
Overall Officials: Contact Lilly at 1-800-LillyRx (1-800-545-5979), Study Director — Eli Lilly and Company
Locations (64):
- United States (34):
  - Cancer Treatment Centers of America, Goodyear, Arizona
  - Mayo Clinic of Scottsdale, Scottsdale, Arizona
  - City of Hope National Medical Center, Duarte, California
  - UCLA Medical Center, Los Angeles, California
  - Kaiser Permanente, Oakland, California
  - Irvine Medical Center, Orange, California
  - University of California - San Diego, San Diego, California
  - Univ of California San Francisco, San Francisco, California
  - Kaiser Permanente, Santa Clara, California
  - Kaiser Permanente Medical Center, Vallejo, California
  - Memorial Cancer Institute, Hollywood, Florida
  - Mayo Clinic in Florida, Jacksonville, Florida
  - Florida Hospital, Orlando, Florida
  - Tallahassee Memorial Cancer Center, Tallahassee, Florida
  - University Cancer and Blood Center, Athens, Georgia
  - Emory University, Atlanta, Georgia
  - University of Chicago Medicine-Comprehensive Cancer Center, Chicago, Illinois
  - Cancer Treatment Centers of America, Zion, Illinois
  - Massachusetts General Hospital, Boston, Massachusetts
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - University of Michigan, Ann Arbor, Michigan
  - START Midwest, Grand Rapids, Michigan
  - Mayo Clinic, Rochester, Minnesota
  - Comprehensive Cancer Centers of Nevada, Las Vegas, Nevada
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - Cleveland Clinic Foundation, Cleveland, Ohio
  - Ohio State University Medical Center, Columbus, Ohio
  - Cancer Treatment Centers of America, Tulsa, Oklahoma
  - University of Pennsylvania Hospital, Philadelphia, Pennsylvania
  - Eastern Regional Medical Center, Philadelphia, Pennsylvania
  - Oncology Consultants, Houston, Texas
  - University of Texas MD Anderson Cancer Center, Houston, Texas
  - Virginia Cancer Specialists, Fairfax, Virginia
  - University of Wisconsin-Madison Hospital and Health Clinic, Madison, Wisconsin
- Australia (5):
  - NSW Health - Sydney Local Health District, Camperdown, New South Wales
  - Royal North Shore Hospital, St Leonards, New South Wales
  - Queensland Health - Metro North Hospital and Health Service, Chermside, Queensland
  - Peter MacCallum Cancer Centre, Melbourne, Victoria
  - Linear Clinical Research, Nedlands, Western Australia
- France (3):
  - Institut Bergonié - Centre Régional de Lutte Contre Le Cancer de Bordeaux et Sud Ouest, Bordeaux, Aquitaine
  - AP-HM, Marseille
  - Gustave Roussy, Villejuif
- Germany (3):
  - Universitätsklinikum Würzburg A. ö. R., Würzburg, Bavaria
  - Universitätsklinikum Köln, Cologne, North Rhine-Westphalia
  - Charité Campus Virchow-Klinikum, Berlin
- Prince of Wales Hospital, Hong Kong, Shatin, New Territories, Hong Kong
- Israel (3):
  - Sheba Medical Center, Ramat Gan, Central District
  - Shaare Zedek Medical Center, Jerusalem, Jerusalem
  - Soroka Medical Center - Pediatric Outpatient Clinic, Beersheba
- Italy (2):
  - Istituto Nazionale dei Tumori, Milan, Lombardy
  - Azienda Ospedaliero Universitaria Pisana, Pisa, PI
- Japan (6):
  - National Cancer Center Hospital East, Kashiwa, Chiba
  - Hokkaido University Hospital, Sapporo, Hokkaido
  - Kanazawa University Hospital, Kanazawa, Ishikawa-ken
  - National Cancer Center Hospital, Chuo-ku, Tokyo
  - Tottori University Hospital, Yonago, Tottori
  - Osaka City General Hospital, Osaka
- University of Auckland, Auckland, New Zealand
- Poland (2):
  - Uniwersyteckie Centrum Kliniczne, Gdansk
  - Centrum Onkologii Instytut im Marii Curie w Warszawie, Warsaw
- National Cancer Centre Singapore, Singapore, Central Singapore, Singapore
- Spain (2):
  - Hospital Universitari Vall d'Hebron, Barcelona, Barcelona [Barcelona]
  - Hospital Madrid Norte Sanchinarro, Madrid
- Kantonsspital Luzern, Lucerne, Canton of Lucerne, Switzerland

REFERENCES:
- [Derived] Rotow J, Patel JD, Hanley MP, Yu H, Awad M, Goldman JW, Nechushtan H, Scheffler M, Kuo CS, Rajappa S, Harada G, Clifford S, Santucci A, Silva L, Tupper R, Oxnard GR, Kherani J, Drilon A. Osimertinib and Selpercatinib Efficacy, Safety, and Resistance in a Multicenter, Prospectively Treated Cohort of EGFR-Mutant and RET Fusion-Positive Lung Cancers. Clin Cancer Res. 2023 Aug 15;29(16):2979-2987. doi: 10.1158/1078-0432.CCR-22-2189. PMID 36996322
- [Derived] Murciano-Goroff YR, Falcon CJ, Lin ST, Chacko C, Grimaldi G, Liu D, Wilhelm C, Iasonos A, Drilon A. Central Nervous System Disease in Patients With RET Fusion-Positive NSCLC Treated With Selpercatinib. J Thorac Oncol. 2023 May;18(5):620-627. doi: 10.1016/j.jtho.2023.01.008. Epub 2023 Jan 16. PMID 36657661